CLINICAL TRIAL: NCT01259791
Title: Evaluation of Patients With Statin Myopathy Using an N of 1 Trial Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Tisha Joy, Assistant Professor, Division of Endocrinology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R-10-450; 17352 (Other: Office of Research Ethics, UWO)
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Statin Myopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Statin (Experimental): Individual-specific statin causing myopathy - i.e., Patients will receive the specific statin previously associated with myopathic symptoms in them (can be any of the following statins: rosuvastatin, atorvastatin, simvastatin, fluvastatin, pravastatin in any of the doses causing symptoms previously).
  Interventions: Drug: Individual-specific statin causing myopathy
- Placebo (Placebo Comparator): Identical placebo to patient-specific statin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Individual-specific statin causing myopathy — Individual-specific statin causing myopathy vs. placebo
  Arms: Statin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study consists of a series of prospective, randomized placebo-controlled n of 1 trials to objectively evaluate the reproducibility of subjective and objective symptoms among patients with a history of statin-related myopathy.

ELIGIBILITY:
Inclusion Criteria:

* history of muscle symptoms occuring within 3 weeks of starting a statin
* need for statin therapy to achieve LDL target according to the 2009 Canadian Lipid Guidelines
* willingness to re-try statin therapy

Exclusion Criteria:

* currently tolerant of statin therapy
* metabolic or inflammatory myopathy
* known neuropathy
* CK elevation >3 times upper limit of normal (ULN) previously on a statin or history of rhabdomyolysis
* pregnant, breastfeeding, or wanting to become pregnant in the near future
* participation in another clinical trial
* other medical condition associated with decreased life span
* inability to adhere to stringent regimen
* unwilling to stop consumption of grapefruit juice

Subset of 5 patients also completing neuromuscular testing:

Inclusion Criteria:

- same as above

Exclusion Criteria:

* same as above but also:
* angina III of IV
* decompensated heart failure
* history of orthopedic problems
* have any skin ulcers or other non-healed skin areas or infections in the arm or leg

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To assess the reliability and reproducibility of subjective symptoms of myalgias to active statin therapy. | Duration of study September 2010 to August 2013

SECONDARY OUTCOMES:
To delineate the relation of objective changes in non-invasive neuromuscular testing to subjective symptoms during the first exposure to active or placebo therapy, in subset of 5 patients with prior history of statin myopathy. | September 2010 to August 2013

CONTACTS AND LOCATIONS:
Overall Officials: Tisha Joy, MD, FRCPC, Principal Investigator — St. Joseph's Health Care, UWO
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Derived] Joy TR, Monjed A, Zou GY, Hegele RA, McDonald CG, Mahon JL. N-of-1 (single-patient) trials for statin-related myalgia. Ann Intern Med. 2014 Mar 4;160(5):301-10. doi: 10.7326/M13-1921. PMID 24737272